CLINICAL TRIAL: NCT06068647
Title: Synergistic Assessment of Ultrasound Data and Respiratory physiOlogical Signals in luNg Diseases
Brief Title: Ultrasound and Respiratory Physiological Signals in Lung Diseases
Acronym: SAURON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Onera BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID4710
Record Dates: First submitted 2023-06-05; First posted 2023-10-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Disease; Interstitial Lung Diseases; Interstitial Pneumonia; Chronic Obstructive Pulmonary Disease; Emphysema or COPD; Ultrasonography; Ultrasound Imaging; Ultrasound
Keywords: Ultrasound; Ultrasound Imaging; Ultrasonography; Emphysema; Chronic obstructive pulmonary disease; Interstitial pneumonia; Interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thoracic ultrasonographic, tomographic and patch-based cardio-respiratory evaluations (Experimental): Ultrasonographic findings will be obtained with clinical machines. Additionally, ultrasonographic scans as acquired with research platform will also be gathered. Metal cutaneous landmarks will be positioned and left during computed tomography scans, indicating the areas of ultrasonographic assessment. This method will support a more accurate comparison between ultrasonographic patterns and CT scans peripheral lung findings.
  Finally, on the same day of enrolment, a wearable system for measuring physiological signals, will be applied. The sensors will be applied to the upper chest. The following information will be collected by each sensor: ECG, respiratory effort, respiratory flow, activity, position, and sound pressure level.
  Interventions: Diagnostic Test: Lung ultrasound, computed tomographic scan and patch-based cardio-respiratory evaluations

INTERVENTIONS:
Diagnostic Test: Lung ultrasound, computed tomographic scan and patch-based cardio-respiratory evaluations — Ultrasonographic findings will be obtained with machines supplied with clinical Units. Additionally, US scans as acquired with open research platform will also be gathered. For both scanners, ultrasonographic scans will be performed and videos will be recorded and stored in each landmark. Metal cutaneous landmarks will be positioned and left during computed tomographic (CT) scans, indicating the areas of ultrasonographic assessment.
  Finally, on the same day of enrolment, a wearable system for measuring physiological signals, will be applied. Within the scope of this study, sensors will be applied to the upper chest. The following information will be collected by each sensor: electrocardiography, respiratory effort, respiratory flow, activity, position, and sound pressure level.

SUMMARY:
The use of lung ultrasound is instrumental in the evaluation of many chest pathologies and its ability to detect pleuro-pulmonary pathology is widely accepted.

However, the use of ultrasound to explore the state of the peripheral lung parenchyma, when the organ is still aerated, is a relatively new application.

Horizontal and vertical artifacts are separate and distinct artifacts that can be seen during ultrasound examination of the lungs. While the practical role of lung ultrasound artifacts is accepted to detect and monitor many conditions, further research is needed for the physical interpretation of ultrasound artifacts. These artifacts are diagnostic signs, but we don't fully understand their origin.

The artifactual information deriving from the surface acoustic interaction, beyond the pleural line, in the ultrasound images of the normally aerated and non-deflated lung, represents the final result of complex interactions of acoustic waves with a specific three-dimensional structure of the biological tissue. Thus, the umbrella term "vertical artifacts" oversimplifies many physical phenomena associated with a pathological pleural plane. There is growing evidence that vertical artifacts are caused by physiological and pathological changes in the superficial lung parenchyma.

Therefore, the need emerges to explore the physical phenomena underlying the artifactual ultrasound information deriving from the surface acoustic interaction of ultrasound with the pleuro-pulmonary structures.

DETAILED DESCRIPTION:
In the last years, lung ultrasonography has gained ever-growing clinical interest and curiosity because of its peculiar ability to acquire clinical information at bedside, its non-invasiveness and low cost. In particular settings (emergency medicine, intensive care unit) its utility has been well demonstrated.

Clinicians use chest ultrasound for detecting pleural diseases, consolidations, bronchiolitis, interstitial lung pathology and critical pulmonary conditions of adults, children, and infants.

However, the development of lung ultrasonography for exploring non-consolidated organs, has been not supported by a strong knowledge of the physical mechanisms that underlie pulmonary artifacts.

Lung ultrasonography is comparable to a standard morphological sonography only when assessing a pulmonary consolidation, a tissue without air, which is in direct contact with the visceral pleural. In this case, the clinicians evaluate anatomic images, representing the real structure of the diseased organ. Differently, when the lung surface is denser but not yet consolidated, the large acoustic impedance gradient between the chest wall and the pulmonary tissue containing air prevents every anatomic representation, and the scan results in the visualization of many kinds of vertical artifacts known as B-Lines.

Even though the practical role of lung ultrasound artifacts is accepted for detecting and monitoring many conditions, many of the published studies are empirical and further research is needed to clarify the physical genesis of vertical artifacts. These artifacts are diagnostic signs, but we do not fully understand their origin. The artifactual information beyond the pleura line in ultrasonographic images of the normal and of the not critically deflated lung represents the ultimate outcome of complex interactions of a specific acoustic wave with a specific three-dimensional structure of the biological tissue.

There is growing evidence that vertical artifacts are caused by physiological and pathological changes in the superficial lung parenchyma.

The study intends to explore the relationship among ultrasound, tomographic and patch-based cardio-respiratory data, obtained from a heterogeneous population of patients suffering from: 1) pre-consolidative pulmonary changes such as diffuse interstitial lung diseases during exacerbation, 2) infectious interstitial pneumonia and 3) chronic obstructive pulmonary disease during both stable phase and exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* inpatients admitted to the hospital due to diffuse interstitial lung diseases during exacerbation OR infectious interstitial pneumonia not caused by SARS-CoV-2 OR acute exacerbation of chronic obstructive pulmonary disease.
* Outpatients with pulmonary paraseptal and/or panlobular emphysema and/or chronic obstructive pulmonary disease during stable phase.
* Patients able to give written informed consent.

Exclusion Criteria:

* history of skin irritation, redness, itching or allergic cutaneous symptoms.
* Allergic reactions to adhesives or hydrogels.
* Family history of adhesive skin allergies.
* Presence of severe skin conditions such as wounds, burns or on any damaged skin.
* Presence of strong magnetic fields in the study setting.
* Presence of electromagnetic disturbances or significant ionizing radiation sources which might lead to signal artifacts.
* Use of external cardiac defibrillators.
* Use of diaphragmatic pacers.
* Use of extra cardiac stimulators.
* Pregnancy.
* Pediatric population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evidence of lung parenchymal involvement evaluated by lung ultrasound. | At enrollment.
  Ultrasonographic findings will be characterized according to internationally recognized and standardized score (LUS COVID protocol, doi:10.1002/jum.15285). Scoring procedures include: score 0 (the pleural line is continuous and regular; horizontal artifacts are present); score 1 (the pleural line is indented. Below the indent, vertical areas of white are visible); score 2 (the pleural line is broken. Below the breaking point, small-to-large, consolidated areas appear with associated areas of white below the consolidated area; score 3 (dense and extended white lung with or without larger consolidations).
Evidence of paraseptal and/or panlobular emphysema. | At enrollment.
  Computed tomographic evidence of paraseptal and/or panlobular emphysema.
Evidence of computed tomographic features and patterns of interstitial lung diseases. | At enrollment.
  Evidence of following features: 1) the presence or absence of pulmonary fibrosis 2) HRCT patterns of reticulation, honeycombing, ground glass and emphysema, as defined in the Fleischner society glossary of thoracic imaging (doi: 10.1148/radiol.2462070712) and 3) severity of traction bronchiectasis.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Inchingolo, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS; Andrea Smargiassi, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soldati G, Demi M, Inchingolo R, Smargiassi A, Demi L. On the Physical Basis of Pulmonary Sonographic Interstitial Syndrome. J Ultrasound Med. 2016 Oct;35(10):2075-86. doi: 10.7863/ultra.15.08023. Epub 2016 Aug 8. No abstract available. PMID 27503755
- [Background] Mento F, Khan U, Faita F, Smargiassi A, Inchingolo R, Perrone T, Demi L. State of the Art in Lung Ultrasound, Shifting from Qualitative to Quantitative Analyses. Ultrasound Med Biol. 2022 Dec;48(12):2398-2416. doi: 10.1016/j.ultrasmedbio.2022.07.007. Epub 2022 Sep 23. PMID 36155147
- [Background] Mento F, Soldati G, Prediletto R, Demi M, Demi L. Quantitative Lung Ultrasound Spectroscopy Applied to the Diagnosis of Pulmonary Fibrosis: The First Clinical Study. IEEE Trans Ultrason Ferroelectr Freq Control. 2020 Nov;67(11):2265-2273. doi: 10.1109/TUFFC.2020.3012289. Epub 2020 Jul 27. PMID 32746228
- [Background] Demi L, van Hoeve W, van Sloun RJG, Soldati G, Demi M. Determination of a potential quantitative measure of the state of the lung using lung ultrasound spectroscopy. Sci Rep. 2017 Oct 6;7(1):12746. doi: 10.1038/s41598-017-13078-9. PMID 28986558
- [Background] Demi L, Demi M, Prediletto R, Soldati G. Real-time multi-frequency ultrasound imaging for quantitative lung ultrasound - first clinical results. J Acoust Soc Am. 2020 Aug;148(2):998. doi: 10.1121/10.0001723. PMID 32872996
- [Background] Soldati G, Inchingolo R, Smargiassi A, Sher S, Nenna R, Inchingolo CD, Valente S. Ex vivo lung sonography: morphologic-ultrasound relationship. Ultrasound Med Biol. 2012 Jul;38(7):1169-79. doi: 10.1016/j.ultrasmedbio.2012.03.001. Epub 2012 May 12. PMID 22579543
- [Background] Smargiassi A, Inchingolo R, Soldati G, Copetti R, Marchetti G, Zanforlin A, Giannuzzi R, Testa A, Nardini S, Valente S. The role of chest ultrasonography in the management of respiratory diseases: document II. Multidiscip Respir Med. 2013 Aug 9;8(1):55. doi: 10.1186/2049-6958-8-55. PMID 23937897
- [Background] Soldati G, Demi M, Smargiassi A, Inchingolo R, Demi L. The role of ultrasound lung artifacts in the diagnosis of respiratory diseases. Expert Rev Respir Med. 2019 Feb;13(2):163-172. doi: 10.1080/17476348.2019.1565997. Epub 2019 Jan 10. PMID 30616416